CLINICAL TRIAL: NCT07375615
Title: Hypoglycemia and Continuous Glucose Monitoring in Neonates (Continuous Sweet Babies Study - CSBS I)
Brief Title: Continous Glucose Monitoring in Neonates at Risk of Hypoglycaemia- a Feasibility Study
Acronym: CSBS I
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: 2022101a
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hyperglycemia; Hypoglycemia; Hypoglycemia Neonatal
Keywords: Neonate, glucose, hypoglycemia, Continous glucose measurement (CGM),newborn
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodsamples analyzed in bloodgasmachine for glucose values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Neonates at risk of hypoglycemia after birth: CGM sensor placed on infant as soon as possible after birth, taken off after 72 hrs, 2 bloodspecimens drawn from babies at different timepoints to compare with CGM values. CGM used to describe glucose profile variation.
  Interventions: Device: Continous glucose monitor

INTERVENTIONS:
Device: Continous glucose monitor — Aplication of CGM device on neonates upper tigh

SUMMARY:
The study's main purpose is to test feasibility of Continous Glucose montoring in Neonates during the first 72 hrs.

DETAILED DESCRIPTION:
The overall aim of this study is to compare and evaluate the feasibility and effectiveness of CGM in clinical care of neonates and increase knowledge of hypoglycemia and neonatal glucose values.

Hypotheses: * CGM detects neonatal hypoglycemia by rapid response to changes in blood glucose levels more effectively than repeated capillary blood sampling

* CGM accurately reflects blood glucose levels within the range relevant for newborn infants. * CGM is safe and easily applied to newborn infants and allows real-time monitoring of tissue glucose levels.

Objective: Examine the feasibility of CGM-device with blood glucose assessments in neonates at risk of hypoglycemia.

• Primary outcome: Hypoglycemic episodes (glucose < 2.6 mmol/L) and rapid changes in glucose values not detected by capillary blood sampling.

Recruitment

• ForCSBSI, recruitment of participants will be carried out at the maternity outpatient clinic at SIHF Lillehammer. In Innlandet Hospital Trust, the vast majority of pregnant women with risk factors of neonatal hypoglycemia are selected for delivery at Lillehammer hospital.

Due to only one sensor available we decided to include 25 neonates in order to test feasibility in a clinical setting.

The CGM-sensor will be applied on the lateral side of the upper thigh within 1 hour after birth. Doctors, midwives and nurses at the maternity ward will be trained in application of the devices and supervision will be offered throughout the entire project whenever requested. Capillary blood glucose measurements, enteral nutrition and other treatments and interventions will follow the standard guideline and procedure recommended by the Norwegian Neonatology Interest group. Exact time points for blood sampling will be registered by the nurse, midwife or parent in a registration form specially designed. Continuous glucose values will be sampled for up to 72 hours. Data will be downloaded from the CGM device storage solution and stored in a secure database. The sensor value will be blinded during sampling time. The neonates will be treated after existing guidelines and all treatment interventions based on standard capillary blood samples. Data from the CGM-devices and capillary blood samples will be analyzed and compared retrospectively.

Sampling and registration of data Capillary blood samples will be analyzed with radiometer technique. Validation will be secured through the ISO-recommendation. Sampling technique will be secured ahead of the project.

Due to the nature of the study and research ethics, the results will be unblinded and episodes of incidentally detected hypoglycemia will be treated according to national guidelines.

The neonate will be monitored for up to 72 hours. Variations in glucose, including rapid drops registered by the CGM-devices will be assessed. This will answer if CGM-sensors have clinically acceptable feasibility in neonates at risk of hypoglycemia, and if episodes of hypoglycemia can be detected earlier with CGM. The nurse or midwife responsible for the baby while admitted to the maternity ward or NICU will be asked to a few questions on clinical observations of symptoms. This will answer if the CGM-sensors are able to detect asymptomatic episodes of hypoglycemia in need of treatment. Number of neonates with registered hypoglycemias, total number of hypoglycemias as well as median and ranges of hypoglycemic values will be assessed. Frequencies of registered hypoglycemic episodes registered will be compared between CGM-devices and blood glucose by suitable statistical methods. Regression analyses will be used to calculate risks of developing hypoglycemia according to CGM or blood glucose testing adjusting for relevant background variables including birth weight, gender, gestational age, risk group for hypoglycemia. Agreement between CGM and blood glucose values will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* LGA, Maternal diabetes (TID and TIID and Gestational diabetes)
* GA>36+6

Exclusion Criteria:

* SGA, Prematurity, major congenital anomalies, multiple pregnancy and severe asphyxia (Apgar < 5 by 10 min. age).

Ages: 0 Hours to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn babies first 72-100Hrs of life
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Glucose profile | +100hrs
  CGM values by sensor compared with Realtime golden standard bloodgas glucose values.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Helge Froisland, MD, PhD, Study Chair — Inland Norway University of Applied Sciences
Locations (1):
- Innlandet hospital trust Lillehammer, Lillehammer, Innlandet, Norway

IPD SHARING:
Plan to Share IPD: No
Regional Ethical board of Norway prohibit sharing individual data on participants in clininical studies this is similar for all studies bot anonymized data and de-identificed data.